CLINICAL TRIAL: NCT03828643
Title: Secukinumab Efficacy Without the Initial Loading Dose at Weeks 0, 1, 2, 3 and 4 in Patients With Chronic Plaque Psoriasis
Brief Title: Secukinumab Efficacy Without the Initial Loading Dose in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Paolo Gisondi, Professor, Universita di Verona
Other Study IDs: Gisondi 3
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis Vulgaris
Keywords: Secukinumab; loading dose; chronic plaque psoriasis; no loading dose
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Cases received secukinumab at the dose 300 mg every 4 weeks from the beginning.
  Interventions: Drug: Secukinumab
- Controls: Controls received secukinumab at the dose 300 mg with loading dose at weeks 0, 1, 2, 3 and 4, followed by monthly maintenance dosing.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300 mg without loading dose at weeks 0, 1, 2, 3 and 4.
  Groups: Cases
Drug: Secukinumab — Secukinumab 300 mg with loading dose at weeks 0, 1, 2, 3 and 4.
  Groups: Controls

SUMMARY:
This was a retrospective, observational study. The objective of the study is investigate the efficacy and safety of secukinumab without the initial weekly loading dose in patients with chronic plaque psoriasis. Patients were stratified in two groups, those receiving secukinumab at the dose 300 mg every 4 weeks from the beginning (cases) and those who received the initial label, weekly loading dose (controls). Efficacy was evaluated by comparing the proportion of patients achieving PASI75 responses at week 16, 32 and 48 between cases and controls. Safety was evaluated by reporting every adverse events up to week 48.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients with moderate to severe chronic plaque psoriasis treated with secukinumab with or without initial loading dose for at least 48 week
* The criteria for receiving secukinumab were according to standard clinical practice.

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with only psoriatic arthritis or with other forms of psoriasis than chronic plaque type (such as drug-induced psoriasis or guttate, erythrodermic, or pustular psoriasis)
* Pregnant women and women during breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe chronic plaque psoriasis attended two Dermatological centers of North Italy in Veneto (Azienda Ospedaliera Universitaria of Verona and Azienda Ospedaliera of Padua) dedicated to the care of patients with psoriasis
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
PASI75 | week 48

SECONDARY OUTCOMES:
PASI90 | week 48

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided